CLINICAL TRIAL: NCT06286553
Title: Trunk Stabilization Exercise and Inspiratory Muscle Training Effects on Diastasis Recti Abdominis in Postpartum Women - A Randomized Controlled Trial
Brief Title: Rehabilitation of Abdominal Diastasis After Childbirth: Trunk and Inspiratory Muscle Training
Acronym: DR-TIME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Patras (Other)
Responsible Party: Principal Investigator, Anastasia Skoura, PhD candidate, University of Patras
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DRA Rehab TEG & IMT
Record Dates: First submitted 2024-02-14; First posted 2024-02-29 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Diastasis Recti And Weakness Of The Linea Alba; Diastasis, Muscle
Keywords: Rehabilitation Research; Telerehabilitation; Exercise Therapy; Breathing Exercise
MeSH Terms: conditions — Diastasis Recti And Weakness Of The Linea Alba; Diastasis, Muscle | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: In this interventional study, three distinct groups are included. The Trunk Exercise Group (TEG) will partake in a comprehensive 12-week therapeutic exercise program that involves progressive strengthening exercises specifically targeting the trunk and pelvic floor muscles, alongside functional retraining exercises. The Trunk Exercise and Inspiratory Muscle Training Group (IMT+TEG) will adhere to the same 12-week therapeutic exercise program as TEG, with additional exercises focusing on strengthening the inspiratory muscles using inspiratory resistance (IMT). The control group (CG) will not participate in the 12-week exercise program but will receive a single exercise session and general management information (oral and written) for DRA.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Trunk Exercise and Inspiratory Muscle Training Group (IMT+TEG) (Experimental): The Trunk Exercise and Inspiratory Muscle Training Group (IMT+TEG) will follow a comprehensive, 12-week therapeutic exercise program that involves progressive strengthening exercises specifically targeting the trunk and pelvic floor muscles, functional retraining exercises, and additional exercises focusing on strengthening the inspiratory muscles (Inspiratory Muscle Training - IMT).
  Interventions: Behavioral: Trunk exercise; Behavioral: Inspiratory Muscle Training (IMT)
- Trunk Exercise Group (TEG) (Active Comparator): The Trunk Exercise Group (TEG) will partake in a comprehensive 12-week therapeutic exercise program that involves progressive strengthening exercises specifically targeting the trunk and pelvic floor muscles, alongside functional retraining exercises.
  Interventions: Behavioral: Trunk exercise
- Control group (CG) (Active Comparator): The control group (CG) will receive general management information for DRA, and written instructions for engaging the deeper abdominals and pelvic floor muscles, accompanied by an educational exercise session. Participants will be encouraged to perform these contractions regularly, without guidance or supervision.
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: Trunk exercise — Trunk stabilization exercises including the following components: (a) progressive deep abdominal muscle retraining (transversus abdominis), (b) progressive pelvic floor muscle retraining, (c) abdominal muscle strengthening exercises (rectus abdominis and obliques), (d) combination of abdominal muscle control and distal extremity movements, and (e) progressive functional exercises.
  Arms: Trunk Exercise Group (TEG); Trunk Exercise and Inspiratory Muscle Training Group (IMT+TEG)
Behavioral: Inspiratory Muscle Training (IMT) — Inspiratory muscle strengthening exercises using inspiratory resistance (IMT devices)
  Arms: Trunk Exercise and Inspiratory Muscle Training Group (IMT+TEG)
Behavioral: Control Group — Participants in the Control Group will receive general management information for DRA, written instructions and a single educational exercise session for contracting the deeper abdominals and pelvic floor muscles.
  Arms: Control group (CG)

SUMMARY:
Diastasis Recti Abdominis (DRA) is the separation of the rectus muscles caused by stretching and thinning of the linea alba during pregnancy and childbirth. It's a common condition, affecting 66-100% of women post-birth and can persist for many years, leading to abdominal protrusion, discomfort, and aesthetic concerns. It might also contribute to back pain, urinary issues, and reduced abdominal strength, impacting quality of life. Recent guidelines propose that conservative management, such as rehabilitation interventions, should be prioritized for DRA. However, there is a lack of consensus among researchers regarding the most effective exercise regimen, resulting in diverse rehabilitation programs. Recent evidence advocates not only for closing the gap but also for achieving optimal function. Current studies often neglect to address functional rehabilitation, underscoring the necessity for robust clinical trials, which is the primary focus of this study.

Additionally, although breathing exercises are commonly prescribed for DRA, the precise role of the diaphragm, the primary respiratory muscle, in rehabilitation hasn't been fully examined. The diaphragm forms the upper boundary of the abdominal cavity and plays a key role in the stability of the trunk, working together with the abdominal and pelvic floor muscles. A recent study found reduced diaphragm excursion in postpartum women with lumbopelvic pain during a low postural demanding task, while previous studies suggest that diaphragm training could alleviate such symptoms influencing factors such as diaphragm thickness and excursion, which may be linked to improved trunk stability. Hence, training the diaphragm and accessory inspiratory muscles through Inspiratory Muscle Training (IMT) could potentially play a crucial role in managing DRA.

In summary, the goal of this study is to develop and assess a comprehensive rehabilitation program aimed at effectively reducing DRA and addressing associated dysfunctions. The program will integrate evidence-based rehabilitation interventions, such as trunk stabilization exercises and IMT, targeting all related dysfunctions caused by DRA, and introducing a novel therapeutic protocol not previously implemented. The study will take the form of a prospective, randomized controlled trial (RCT).

DETAILED DESCRIPTION:
The primary objective of the study is to develop and assess a comprehensive rehabilitation program for Diastasis Recti Abdominis (DRA) and associated dysfunctions, through a prospective randomized controlled trial (RCT). The study is aimed at (a) implementing exercise of the superficial and deep abdominal muscles in both concentric and eccentric contractions targeting muscle strength, development, and arrangement of muscle fibers, potentially facilitating the closure of DRA , as well as pelvic floor muscle exercises with adequate loading and progression aiming for optimal muscular adaptations, (b) integrating exercises strengthening the diaphragm and accessory inspiratory muscles (Inspiratory Muscle Training - IMT), to improve diaphragm function (thickness, mobility/excursion) and contribute to the overall optimal function of the trunk, facilitating force transfer through the abdominal wall, especially when combined with exercises tensing the linea alba (transversus abdominis and pelvic floor muscle exercises), (c) progressing simple contraction exercises into functional, according to loading and progression principles for optimal function in static and dynamic conditions, and (d) developing a flexible exercise program that can also be accessed remotely, aiming to enhance women's access to rehabilitation services, potentially enhancing compliance as well.

The study adheres to ethical considerations and the Helsinki Declaration and is approved by the Research Ethics Committee (R.E.C.) of the University of Patras (internal code: 16192/18-12-2023). All participants will be thoroughly informed about the procedure and will be invited to complete the consent form after receiving complete written information about the study and the protection of their data. All patient data will be stored anonymously/coded in a secure cloud platform accessed only by the research team members. Imputation methods will be applied to address situations where variables are missing, uninterpretable, or inconsistent. Any adverse events will be addressed and documented, while medical consultation will be accessible during patient assessment/rehabilitation hours. Any modifications to the study protocol, data collection methods, or other aspects of the study will be reviewed thoroughly among researchers and the Internal Review Board of the R.E.C., and the study protocol as well as study registration will be adjusted accordingly. The accuracy, completeness, and representativeness of registry data is assured by the research team. A comprehensive data dictionary is established among the research team, containing detailed variable descriptions, coding information, and normal ranges, ensuring consistency and clarity in data collection.

Sample recruitment will be through leaflets and posters placed in various areas of the University campus, the University General Hospital of Patras, and the wider region of Achaia, as well as publicizing this research in professional associations (Panhellenic Medical Association, Panhellenic Physiotherapists' Association) and healthcare professionals (obstetricians, gynecologists, urologists, surgeons, etc.) who may encounter such cases. Additionally, informational events will be planned in various areas of Achaia for the general public, and the study will also be promoted on the university website (Department of Physiotherapy webpage), social media, and conferences. Based on the power analysis conducted using GPowerSoftware 3.1.9.7, considering previous studies of good methodological quality and the same primary outcome, a power of 95%, effect size of 0.30, and a significance level of 5% were established. Including an expected dropout rate of up to 20% of the total sample, a total of 48 women are required (39 according to GPowerSoftware plus an additional 20% for possible dropouts). Consequently, each group is estimated to include 16-20 women.

The allocation of participants into different intervention groups (TEG, IMT+TEG, or CG) will be done by a researcher "blinded" to the interventions and assessment methods, using block randomization, creating a sequence of random numbers through specific software. Each participant will be randomly assigned a number from this sequence through a sealed, opaque envelope. Then participants will be randomly allocated to the intervention groups via sealed, opaque envelopes. To ensure homogeneous distribution of the sample among the intervention groups, each block will contain equal number of envelopes for each intervention group. This method ensures both randomization and concealment of allocation, maintaining the integrity and unbiased distribution of the sample. Due to the nature of the treatment, clinicians cannot be "blinded" to the intervention. However, the analysis of the data will be 'blind' (blind assessor). Analysis will be based on data resulting from the initial grouping of patients by treatment protocol (intention-to-treat analysis).

Both assessment and intervention will take place at the Physiotherapy Department of the University of Patras, in the Clinical Physiotherapy and Research Laboratory (CPRlab). Primary outcome measures will be inter-recti distance (IRD), assessed using diagnostic ultrasound (Versana Active™, GE Healthcare, Illinois, US). Secondary outcome measures will include: a) diaphragmatic thickness (inspiratory & expiratory) and excursion measured via diagnostic ultrasound (Versana Active™, GE Healthcare, Illinois, US), b) strength of the inspiratory muscles (measured by MIP, S-Index, PIF) assessed using the POWERbreathe KH2 (HaB International Ltd., Warwickshire, United Kingdom), c) Trunk function, assessed through functional motor control tests including trunk flexion, plank, side plank, McGill's trunk flexor endurance test, and d) specific questionnaires: i) Body Image States Scale (BISS), ii) Activity Assessment Scale (AAS), and iii) Hernia-Related Quality-of-Life Survey (HerQLes). Prior to the study, pilot reliability studies of all assessment tools and feasibility pilot studies will be completed.

Ultrasound measurements will be conducted by two experienced physiotherapists specializing in womens' health and musculoskeletal dysfunctions, who are adequately trained by a radiologist specializing in diagnostic ultrasound and by a fellow physiotherapist who is experienced in using these imaging techniques (Rehabilitative Ultrasound Imaging - RUSI) in daily clinical practice. Both of these healthcare professionals will supervise the assessment procedure and resolve any issues that may arise during the measurements and/or individual analyses. Before the measurements, the examiners will train the participants in diaphragmatic breathing, contraction of deep abdominal muscles (drawing-in maneuver), and pelvic floor muscles (PFM). Women who demonstrate satisfactory control of these muscles will take part in the intervention. Women will also be asked questions regarding their demographics (age, height/weight, etc.), physical condition, and health history. They will subsequently complete the Australian Pelvic Floor Questionnaire (APFQ-GR), which includes questions about bladder and bowel function, sexual health, and potential symptoms related to the pelvic floor. Additionally, they will fill out the International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF-GR). In cases where abdominal wall or lower back pain is reported, patients will be asked to rate the intensity of this pain according to the Numeric Pain Rating Scale (NPRS).

Intervention groups (TEG and IMT+TEG) will follow a comprehensive exercise program that will last 12 weeks and will include the following components: (a) progressive exercises for retraining deep abdominal muscles (transversus abdominis), (b) progressive exercises for retraining pelvic floor muscles, (c) abdominal muscle strengthening exercises (rectus abdominis, obliques), (d) combination of abdominal muscle control and distal extremity movements, and (e) progressive functional exercises. Each session will range from 20 to 45 minutes, with a progressive increase in duration over the weeks. Participants will exercise three times a week, with one or two in-person sessions per 2 weeks at our department's laboratory (CPRlab) under the supervision of experienced physiotherapists, and the rest of the sessions conducted via teleconference, either synchronous or asynchronous. The in-person sessions will occur in small groups of patients and will be supervised by experienced physiotherapists who will adjust or modify exercise progression according to the patients' needs. Teleconference sessions will be conducted via Zoom communications platform (Zoom Video Communications, California, US). Session scheduling, patient communication, and coordination will be facilitated through a blended learning platform (Classroom, Google, California, US), which the research team modified accordingly to present a patient-friendly interface containing useful tools such as leaflets, information, educational videos etc. Exercise compliance will be assessed through exercise diaries uploaded on the platform. If a participant misses a scheduled online session, the exercise session will be recorded and uploaded to the platform. Women will be encouraged to repeat the exercise program as many times as desired during the week, beyond the scheduled sessions supervised by a physiotherapist. Successful completion of the program will require supervised attendance at a minimum of two out of three sessions per week (i.e., >70% attendance). The exercise program's progression will focus on increasing sets, repetitions, exercise complexity, load, and overall program duration. Simple equipment will be used, such as mats, resistance bands, dumbbells, towels, and pillows.

Trunk Exercise and Inspiratory Muscle Training Group (IMT+TEG) will also perform breathing exercises using inspiratory muscle training (IMT) for 12 weeks. Women will perform IMT three times per week. One training session will be in-person (either weekly or 1 in two weeks) using the POWERbreathe Classic IMT (HaB International Ltd.,Warwickshire, United Kingdom) device under the supervision of an experienced physiotherapist. The other two sessions will be conducted via teleconference from home (using the same device) to ensure the adequacy of the training load. Inspiratory muscle exercises will be performed at an intensity of 50-80% of maximum inspiratory pressure (MIP) and will last 5-10 minutes. There will be a total of 3 sets with 8-10 repetitions, performed twice per session. Inspiratory resistance will progressively increase at a rate of 2-3cm H2O per week. Remote IMT sessions will be scheduled before the trunk exercise program to prevent potential patient fatigue.

The control group will not participate in the 12-week exercise program, but will receive a single training session, general information on managing DRA, along with written instructions for proper abdominal and pelvic floor muscle contraction.

Statistical Analysis Data collected will be processed and analyzed using the SPSS program (version 28 for Windows IBM, Armonk, NY, USA). Statistical analysis will identify correlations between the studied variables, and repeated measures ANOVA will be used to identify statistically significant differences among sample groups. Effect sizes with 95% confidence intervals will be calculated for each outcome measure. Effect sizes will be considered large if ≥0.8, moderate if ≥0.5 and small if ≥0.2.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 18-50 years
* Diagnosed with diastasis recti abdominis (DRA) with an inter-recti distance (IRD) greater than 2.8 cm
* Beyond 6 months postpartum (preferably within the range of up to 5 years postpartum)

Exclusion Criteria:

* Severe chronic respiratory disease (i.e. COPD, chronic bronchitis, pulmonary emphysema or fibrosis)
* Connective tissue disorders
* Neurological disorders
* Severe musculoskeletal conditions hindering exercise participation (e.g., severe low back pain, sciatica, etc.)
* Previous abdominal surgeries (excluding cesarean section)
* Delivery within the last 6 months
* BMI greater than 30 kg/m²

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 48 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Inter-recti distance (IRD) | IRD is measured at baseline, at 3 months and at 6 months (follow-up assessment).
  Distance between the rectus muscles measured in cm via diagnostic ultrasound (Mota et al., 2018).

SECONDARY OUTCOMES:
Diaphragmatic Thickness | Diaphragmatic Thickness is assessed at baseline, at 3 months and at 6 months from baseline (follow-up assessment).
  Thickness of the diaphragm measured in cm during maximal inspiration and expiration using ultrasound.
Diaphragmatic Excursion | Diaphragmatic excursion is assessed at baseline, at 3 months and at 6 months from baseline (follow-up assessment).
  Mobility of the diaphragm measured in cm during tidal inspiration and expiration using ultrasound.
Maximum Inspiratory Pressure (MIP) | MIP is assessed at baseline, at 3 months and at 6 months from baseline (follow-up assessment).
  Maximum Inspiratory Pressure measured in cmΗ2Ο using POWERbreathe KH2 device
Strength Index (S-Index) | S-Index is assessed at baseline, at 3 months and at 6 months from baseline (follow-up assessment).
  Inspiratory muscle strength index measured in cmΗ2Ο using POWERbreathe KH2 device
Peak Inspiratory Flow (PIF) | PIF is assessed at baseline, at 3 months and at 6 months from baseline (follow-up assessment).
  Peak Inspiratory Flow measured in L/sec using POWERbreathe KH2 device
Trunk flexion test | Trunk flexion test is assessed at baseline, at 4 weeks, at 8 weeks, at 12 weeks (3 months from baseline) and at 6 months from baseline (follow-up assessment).
  Endurance in a trunk flexion position assessed measuring time (in sec) using a stopwatch
Plank test | Plank test is assessed at baseline, at 4 weeks, at 8 weeks, at 12 weeks (3 months from baseline) and at 6 months from baseline (follow-up assessment).
  Endurance in a plank position assessed measuring time (in sec) using a stopwatch
Side plank test | Side plank test is assessed at baseline, at 4 weeks, at 8 weeks, at 12 weeks (3 months from baseline) and at 6 months from baseline (follow-up assessment)
  Endurance in a side plank position assessed measuring time (in sec) using a stopwatch
McGill's trunk flexor endurance test | McGill's trunk flexor endurance test is assessed at baseline, at 4 weeks, at 8 weeks, at 12 weeks (3 months from baseline) and at 6 months from baseline (follow-up assessment)
  Endurance in a trunk flexion position proposed by McGill and assessed measuring time (in sec), using a stopwatch
Body Image States Scale (BISS) | BISS is assessed at baseline, at 3 months and at 6 months from baseline (follow-up assessment) (follow-up assessment).
  Patient-centered questionnaire which assesses body image perception using 6 questions (1-9 points per question).
Activities Assessment Scale (AAS) | AAS is assessed at baseline, at 3 months and at 6 months from baseline (follow-up assessment) (follow-up assessment).
  A patient-centered questionnaire designed to assess difficulty during activities related to the abdominal wall, through 13 questions, with each question scored on a scale of 1 to 5 points. A rating of 1 indicates "no difficulty," and 5 indicates the patient is "not able to do it." An additional option of 8 points is available when the patient "did not do it for other reasons."
Hernia-Related Quality-of-Life Survey (HerQLes) | HerQLes is assessed at baseline, at 3 months and at 6 months from baseline (follow-up assessment).
  A patient-centered survey that evaluates quality of life related to hernia using a set of 12 questions, with each question rated on a scale of 1 ("strongly disagree") to 6 points ("strongly agree").

CONTACTS AND LOCATIONS:
Overall Officials: Evdokia Billis, PhD, Study Director — University of Patras, Department of Physiotherapy
Locations (1):
- Laboratory of Clinical Rehabilitation and Research (CPRlab), University of Patras, Pátrai, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boissonnault JS, Blaschak MJ. Incidence of diastasis recti abdominis during the childbearing year. Phys Ther. 1988 Jul;68(7):1082-6. doi: 10.1093/ptj/68.7.1082. PMID 2968609
- [Background] Candido G, Lo T, Janssen P. Risk factors for diastasis of the recti abdominis. J Assoc Chart Physiother Womens Health 2005;97:49-54.
- [Background] Sperstad JB, Tennfjord MK, Hilde G, Ellstrom-Engh M, Bo K. Diastasis recti abdominis during pregnancy and 12 months after childbirth: prevalence, risk factors and report of lumbopelvic pain. Br J Sports Med. 2016 Sep;50(17):1092-6. doi: 10.1136/bjsports-2016-096065. Epub 2016 Jun 20. PMID 27324871
- [Background] Parker, M. A., Millar, L. A., & Dugan, S. A. (2009). Diastasis Rectus Abdominis and Lumbo-Pelvic Pain and Dysfunction-Are They Related? J Women's Health Phys Ther. 2008;33(2):15 -22.
- [Background] Gunnarsson U, Stark B, Dahlstrand U, Strigard K. Correlation between abdominal rectus diastasis width and abdominal muscle strength. Dig Surg. 2015;32(2):112-6. doi: 10.1159/000371859. Epub 2015 Mar 5. PMID 25766128
- [Background] Benjamin DR, Frawley HC, Shields N, van de Water ATM, Taylor NF. Relationship between diastasis of the rectus abdominis muscle (DRAM) and musculoskeletal dysfunctions, pain and quality of life: a systematic review. Physiotherapy. 2019 Mar;105(1):24-34. doi: 10.1016/j.physio.2018.07.002. Epub 2018 Jul 24. PMID 30217494
- [Background] van de Water AT, Benjamin DR. Measurement methods to assess diastasis of the rectus abdominis muscle (DRAM): A systematic review of their measurement properties and meta-analytic reliability generalisation. Man Ther. 2016 Feb;21:41-53. doi: 10.1016/j.math.2015.09.013. Epub 2015 Oct 3. PMID 26474542
- [Background] Carlstedt A, Bringman S, Egberth M, Emanuelsson P, Olsson A, Petersson U, Palstedt J, Sandblom G, Sjodahl R, Stark B, Strigard K, Tall J, Theodorsson E. Management of diastasis of the rectus abdominis muscles: recommendations for swedish national guidelines. Scand J Surg. 2021 Sep;110(3):452-459. doi: 10.1177/1457496920961000. Epub 2020 Sep 28. PMID 32988320
- [Background] Gluppe S, Engh ME, Bo K. What is the evidence for abdominal and pelvic floor muscle training to treat diastasis recti abdominis postpartum? A systematic review with meta-analysis. Braz J Phys Ther. 2021 Nov-Dec;25(6):664-675. doi: 10.1016/j.bjpt.2021.06.006. Epub 2021 Jul 21. PMID 34391661
- [Background] Berg-Poppe P, Hauer M, Jones C, Munger M, Wethor C. Use of Exercise in the Management of Postpartum Diastasis Recti: A Systematic Review. J Womens Health Phys Therap, 2022; 46(1):p 35-47, DOI: 10.1097/JWH.0000000000000231
- [Background] Dufour, S., Bernard, S.A., Murray-Davis, B., et al. Establishing Expert-Based Recommendations for the Conservative Management of Pregnancy-Related Diastasis Rectus Abdominis: A Delphi Consensus Study. J Womens Health Phys Therap, 2019; 73-81. doi: 10.1097/JWH.0000000000000130
- [Background] Skoura A, Billis E, Papanikolaou DT, Xergia S, Tsarbou C, Tsekoura M, Kortianou E, Maroulis I. Diastasis Recti Abdominis Rehabilitation in the Postpartum Period: A Scoping Review of Current Clinical Practice. Int Urogynecol J. 2024 Mar;35(3):491-520. doi: 10.1007/s00192-024-05727-1. Epub 2024 Feb 10. PMID 38340172
- [Background] Janssens L, McConnell AK, Pijnenburg M, Claeys K, Goossens N, Lysens R, Troosters T, Brumagne S. Inspiratory muscle training affects proprioceptive use and low back pain. Med Sci Sports Exerc. 2015 Jan;47(1):12-9. doi: 10.1249/MSS.0000000000000385. PMID 24870567
- [Background] Finta R, Nagy E, Bender T. The effect of diaphragm training on lumbar stabilizer muscles: a new concept for improving segmental stability in the case of low back pain. J Pain Res. 2018 Nov 28;11:3031-3045. doi: 10.2147/JPR.S181610. eCollection 2018. PMID 30568484
- [Background] Ahmadnezhad L, Yalfani A, Gholami Borujeni B. Inspiratory Muscle Training in Rehabilitation of Low Back Pain: A Randomized Controlled Trial. J Sport Rehabil. 2020 Nov 1;29(8):1151-1158. doi: 10.1123/jsr.2019-0231. Epub 2020 Jan 7. PMID 31910393
- [Background] Oh D, Kim G, Lee W, Shin MM. Effects of inspiratory muscle training on balance ability and abdominal muscle thickness in chronic stroke patients. J Phys Ther Sci. 2016 Jan;28(1):107-11. doi: 10.1589/jpts.28.107. Epub 2016 Jan 30. PMID 26957739
- [Background] Souza H, Rocha T, Pessoa M, Rattes C, Brandao D, Fregonezi G, Campos S, Aliverti A, Dornelas A. Effects of inspiratory muscle training in elderly women on respiratory muscle strength, diaphragm thickness and mobility. J Gerontol A Biol Sci Med Sci. 2014 Dec;69(12):1545-53. doi: 10.1093/gerona/glu182. PMID 25395284
- [Background] Cheng YY, Lin SY, Hsu CY, Fu PK. Respiratory Muscle Training Can Improve Cognition, Lung Function, and Diaphragmatic Thickness Fraction in Male and Non-Obese Patients with Chronic Obstructive Pulmonary Disease: A Prospective Study. J Pers Med. 2022 Mar 16;12(3):475. doi: 10.3390/jpm12030475. PMID 35330474
- [Background] Kocjan J, Gzik-Zroska B, Nowakowska K, Burkacki M, Suchon S, Michnik R, Czyzewski D, Adamek M. Impact of diaphragm function parameters on balance maintenance. PLoS One. 2018 Dec 28;13(12):e0208697. doi: 10.1371/journal.pone.0208697. eCollection 2018. PMID 30592726
- [Background] Lee K, Cho JE, Hwang DY, Lee W. Decreased Respiratory Muscle Function Is Associated with Impaired Trunk Balance among Chronic Stroke Patients: A Cross-sectional Study. Tohoku J Exp Med. 2018 Jun;245(2):79-88. doi: 10.1620/tjem.245.79. PMID 29848898
- [Background] Jiroumaru T, Wachi M, Noguchi S, Ikeya M, Hattori T, Fujitani R, Suzuki M, Tanida S, Shichiri N, Fujikawa T. Is the diaphragm thickness related to gait speed in patients with hemiplegia caused by cerebrovascular accident? J Phys Ther Sci. 2021 Jun;33(6):450-454. doi: 10.1589/jpts.33.450. Epub 2021 Jun 18. PMID 34177107
- [Background] Hortobagyi T, Hill JP, Houmard JA, Fraser DD, Lambert NJ, Israel RG. Adaptive responses to muscle lengthening and shortening in humans. J Appl Physiol (1985). 1996 Mar;80(3):765-72. doi: 10.1152/jappl.1996.80.3.765. PMID 8964735
- [Background] Roig M, O'Brien K, Kirk G, Murray R, McKinnon P, Shadgan B, Reid WD. The effects of eccentric versus concentric resistance training on muscle strength and mass in healthy adults: a systematic review with meta-analysis. Br J Sports Med. 2009 Aug;43(8):556-68. doi: 10.1136/bjsm.2008.051417. Epub 2008 Nov 3. PMID 18981046
- [Background] Ema R, Akagi R, Wakahara T, Kawakami Y. Training-induced changes in architecture of human skeletal muscles: current evidence and unresolved issues. J Phys Fit Sports Med. 2016;5(1):37-4
- [Background] Mota P, Pascoal AG, Carita AI, Bo K. Normal width of the inter-recti distance in pregnant and postpartum primiparous women. Musculoskelet Sci Pract. 2018 Jun;35:34-37. doi: 10.1016/j.msksp.2018.02.004. Epub 2018 Feb 20. PMID 29494833
- [Background] Tuttle LJ, Fasching J, Keller A, et al. Noninvasive Treatment of Postpartum Diastasis Recti Abdominis: A Pilot Study. J Womens Health Phys Therap, 2018;42(2):65-75. doi:10.1097/JWH.0000000000000101
- [Background] Keshwani N, Mathur S, McLean L. The impact of exercise therapy and abdominal binding in the management of diastasis recti abdominis in the early post-partum period: a pilot randomized controlled trial. Physiother Theory Pract. 2021 Sep;37(9):1018-1033. doi: 10.1080/09593985.2019.1675207. Epub 2019 Oct 23. PMID 31642725
- [Background] Boussuges A, Rives S, Finance J, Bregeon F. Assessment of diaphragmatic function by ultrasonography: Current approach and perspectives. World J Clin Cases. 2020 Jun 26;8(12):2408-2424. doi: 10.12998/wjcc.v8.i12.2408. PMID 32607319
- [Background] Silva PE, de Carvalho KL, Frazao M, Maldaner V, Daniel CR, Gomes-Neto M. Assessment of Maximum Dynamic Inspiratory Pressure. Respir Care. 2018 Oct;63(10):1231-1238. doi: 10.4187/respcare.06058. Epub 2018 Jul 17. PMID 30018174
- [Background] Langer D, Jacome C, Charususin N, Scheers H, McConnell A, Decramer M, Gosselink R. Measurement validity of an electronic inspiratory loading device during a loaded breathing task in patients with COPD. Respir Med. 2013 Apr;107(4):633-5. doi: 10.1016/j.rmed.2013.01.020. Epub 2013 Feb 17. PMID 23421970
- [Background] Van Hollebeke M, Poddighe D, Gojevic T, Clerckx B, Muller J, Hermans G, Gosselink R, Langer D. Measurement validity of an electronic training device to assess breathing characteristics during inspiratory muscle training in patients with weaning difficulties. PLoS One. 2021 Aug 26;16(8):e0255431. doi: 10.1371/journal.pone.0255431. eCollection 2021. PMID 34437582
- [Background] Hislop, Helen J. Daniels & Worthingham's Muscle Testing : Techniques of Manual Examination. St. Louis, Mo. :Saunders Elsevier, 2007. APA
- [Background] Kim S, Yi D, Yim J. The Effect of Core Exercise Using Online Videoconferencing Platform and Offline-Based Intervention in Postpartum Woman with Diastasis Recti Abdominis. Int J Environ Res Public Health. 2022 Jun 8;19(12):7031. doi: 10.3390/ijerph19127031. PMID 35742279
- [Background] Cash TF, Fleming EC, Alindogan J, Steadman L, Whitehead A. Beyond body image as a trait: the development and validation of the Body Image States Scale. Eat Disord. 2002 Summer;10(2):103-13. doi: 10.1080/10640260290081678. PMID 16864251
- [Background] McCarthy M Jr, Jonasson O, Chang CH, Pickard AS, Giobbie-Hurder A, Gibbs J, Edelman P, Fitzgibbons R, Neumayer L. Assessment of patient functional status after surgery. J Am Coll Surg. 2005 Aug;201(2):171-8. doi: 10.1016/j.jamcollsurg.2005.03.035. PMID 16038812
- [Background] Krpata DM, Schmotzer BJ, Flocke S, Jin J, Blatnik JA, Ermlich B, Novitsky YW, Rosen MJ. Design and initial implementation of HerQLes: a hernia-related quality-of-life survey to assess abdominal wall function. J Am Coll Surg. 2012 Nov;215(5):635-42. doi: 10.1016/j.jamcollsurg.2012.06.412. Epub 2012 Aug 4. PMID 22867715
- [Background] Billis E, Kritikou S, Konstantinidou E, Fousekis K, Deltsidou A, Sergaki C, Giannitsas K. The Greek version of the Australian Pelvic Floor Questionnaire: Cross-cultural adaptation and validation amongst women with urinary incontinence. Eur J Obstet Gynecol Reprod Biol. 2022 Dec;279:171-175. doi: 10.1016/j.ejogrb.2022.10.025. Epub 2022 Nov 2. PMID 36347115
- [Background] Athanasiou S, Grigoriadis T, Kyriakidou N, Giannoulis G, Antsaklis A. The validation of international consultation on incontinence questionnaires in the Greek language. Neurourol Urodyn. 2012 Sep;31(7):1141-4. doi: 10.1002/nau.22197. Epub 2012 Apr 16. PMID 22508384
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748